CLINICAL TRIAL: NCT00494663
Title: A Phase 2b, Randomized, Double-Blind, Parallel-Group, Study of Safety and Efficacy of 16 Weeks of Treatment With DIO-902 or DIO-902 Placebo in Addition to Metformin and Atorvastatin or Atorvastatin Placebo in Subjects With Type 2 Diabetes Mellitus (Protocol No. DIO-502)
Brief Title: A Phase 2b Study of DIO-902 or DIO-902 Placebo in Addition to Metformin and Atorvastatin or Atorvastatin Placebo for Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Program Terminated
Sponsor: DiObex (Industry)
Responsible Party: Bernice Welles, MD, DiObex, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIO-502
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; type 2 diabetes; cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Experimental): 150mg DIO-902 + 10mg atorvastatin
  Interventions: Drug: DIO-902
- 2 (Experimental): 300mg DIO-902 + 10mg atorvastatin
  Interventions: Drug: DIO-902
- 3 (Experimental): 450mg DIO-902 + 10mg atorvastatin
  Interventions: Drug: DIO-902
- 4 (Placebo Comparator): DIO-902 Placebo + 10mg atorvastatin
  Interventions: Drug: DIO-902 placebo
- 5 (Experimental): 150mg DIO-902 + atorvastatin placebo
  Interventions: Drug: DIO-902
- 6 (Experimental): 300mg DIO-902 + atorvastatin placebo
  Interventions: Drug: DIO-902
- 7 (Experimental): 450mg DIO-902 + atorvastatin placebo
  Interventions: Drug: DIO-902
- 8 (Placebo Comparator): DIO-902 placebo + atorvastatin placebo
  Interventions: Drug: DIO-902 placebo

INTERVENTIONS:
Drug: DIO-902 — 150mg tablet once per day for 16 weeks
  Other Names: 2S,4R enantionmer of ketoconazole
  Arms: 1
Drug: DIO-902 — 300mg tablet once per day for 16 weeks
  Other Names: 2S,4R enantiomer of ketoconazole
  Arms: 2
Drug: DIO-902 — 450mg DIO-902 tablet once daily for 16 weeks
  Other Names: 2S,4R enantiomer of ketoconazole
  Arms: 3
Drug: DIO-902 placebo — DIO-902 placebo tablet once daily for 16 weeks
  Arms: 4
Drug: DIO-902 — 150mg tablet of DIO-902 once daily for 16 weeks
  Other Names: 2S,4R enantiomer of ketoconazole
  Arms: 5
Drug: DIO-902 — 300mg DIO-902 tablet daily for 16 weeks
  Other Names: 2S,4R enantiomer of ketoconazole
  Arms: 6
Drug: DIO-902 — 450mg DIO-902 tablet for 16 weeks
  Other Names: 2S,4R enantiomer of ketoconazole
  Arms: 7
Drug: DIO-902 placebo — DIO-902 placebo tablet once daily for 16 weeks
  Arms: 8

SUMMARY:
DiObex Inc. is developing an experimental drug (DIO-902) that is made up of part of the ketoconazole molecule for the treatment of elevated blood glucose associated with type 2 diabetes mellitus. Ketoconazole (Nizoral®) is a drug available by prescription for the treatment of fungal infections however DIO-902 is an investigational drug. DIO-902 may lower blood glucose by lowering levels of a naturally occurring hormone called cortisol. Elevated cortisol may contribute to the development of type 2 diabetes.

The purpose of this research study is to test the safety of DIO-902 when taken by mouth with metformin and the cholesterol-lowering drug atorvastatin to determine the type and severity of any side effects from this treatment.

Other purposes of the study are to see how the treatment affects your blood glucose levels, cholesterol levels, blood pressure, and waist circumference.

DETAILED DESCRIPTION:
DIO-902 may lower blood glucose by lowering levels of a naturally occurring hormone called cortisol. Elevated cortisol may contribute to the development of type 2 diabetes. Clinical trials with ketoconazole have been carried out in patients with type 2 diabetes. Three clinical trials with DIO-902 have been completed in which 37 patients with type 2 diabetes and 42 normal healthy volunteers (people without type 2 diabetes) were enrolled. Patients in these studies received multiple doses of DIO-902. DIO-902 may reduce the level of cortisol in your blood and therefore may provide you with better control of your blood glucose levels.

STUDY DRUG ASSIGNMENT

You will be randomized, that is, given a 1 in 4 chance of receiving either 150mg/day of DIO-902, 300mg/day of DIO-902, 450mg/day of DIO-902 or DIO-902 placebo and a 1 in 2 chance of receiving 10mg/day of atorvastatin or atorvastatin placebo. The study drug is a tablet and will be taken by mouth with water. You will take 3 tablets of DIO-902 or DIO-902 placebo and 1 tablet of atorvastatin or atorvastatin placebo each day. The tablets will be taken at the same time each day (2200h or 10:00pm). Neither you nor your doctor will know which dose of DIO-902 or DIO-902 placebo you are on or whether you are taking the atorvastatin or atorvastatin placebo. If necessary, your doctor has a way of finding out which dose you were assigned.

Atorvastatin

If you are taking any cholesterol-lowering drugs, these drugs must be discontinued on the day prior to the Pre-Treatment Visit (Week -4) and for the duration of the study. At Visit 1 (Week 0) you will be assigned to DIO-902 or DIO-902 placebo and to either atorvastatin or atorvastatin placebo. You will continue to take the assigned drug until Study Visit 4 (Week 8). At Study Visit 4 (Week 8) all patients will begin taking atorvastatin through the remainder of the study. Your DIO-902 or DIO-902 placebo assignment will remain the same. Atorvastatin tablets will be supplied to you until Study Visit 6 (Week 16). At this visit you will be given a prescription for a 28 day supply of atorvastatin 10mg.day to last until Study Visit 7 (Week 20).

There will a total of 9 study visits. At each visit all or some of the following will occur: blood and urine samples will be taken, physical exam, assessment of side effects, and ECG will be performed.

ELIGIBILITY:
Inclusion Criteria:

-

A subject may be included in this study if he/she meets all of the following criteria:

1. Male or female, age 18 to 75
2. Females of childbearing potential (intact uterus and within 1 year since the last menstrual period) should be non-lactating and have a negative serum pregnancy test. In addition, these subjects should agree to use the following acceptable birth control methods beginning at the Screening Visit and throughout the study:

   1. abstinence
   2. surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum
   3. IUD in place for at least 3 months
   4. barrier methods (condom or diaphragm) with spermicide
   5. surgical sterilization of the partner (vasectomy for 6 months)
   6. hormonal contraceptives for at least 3 months prior to the first dose
3. Diagnosis of type 2 diabetes mellitus (DM) for at least 6 months.
4. Type 2 diabetes may be treated only with metformin (metformin hydrochloride tablets or metformin hydrochloride extended-release tablets) at a total daily dose of 500 mg to the maximum labeled dose. (See Appendix G for List of Drug Trade Names).The dose of metformin must be stable for >8 weeks prior to the Pre-Treatment Visit (Week -4) and throughout the course of the study. The subject must not be on any other pharmacologic or over-the-counter treatments for diabetes.
5. HbA1C level of 7.0 to 10.0%
6. Fasting C-peptide level of >0.33 nmol/l (1.0 ng/ml)
7. ACTH stimulation test results with any cortisol level of >18 µg/dl at baseline or 60 minutes
8. Normal complete blood count (CBC) with platelets and differential
9. 12-lead electrocardiogram (ECG) shows no acute ischemia or clinically significant abnormality. Subjects with QTc interval of >450 msec will be excluded from the study.
10. BMI of 27 to 42 kg/m2 (see Appendix B)
11. Subjects with a history of hypertension may be on a stable anti-hypertensive regimen for (except those drugs stated under Exclusion Criterion 8) for >6 weeks prior to the Pre-Treatment Visit (Week -4))
12. Ability to comprehend and a willingness to provide informed consent

Exclusion Criteria:

* A subject may be excluded from this study if he/she meets any of the following criteria:

  1. Previous participation in a clinical trial with DIO-902.
  2. History of any atherosclerotic disorder (myocardial infarction, unstable angina, cerebrovascular accident, peripheral vascular disease or congestive heart failure secondary to ischemic myocardial injury) that would, in the estimation of the Investigator, make it unsafe to stop all lipid lowering drugs for up to 12 weeks during the course of the study.
  3. Known hypersensitivity or idiosyncratic reaction related to ketoconazole or other imidazole compounds.
  4. History of malignancy (except basal cell carcinoma) within the 3 years before the initial dose of the study medication.
  5. Excessive alcohol intake (>20 g per day for females (1.5 standard alcohol drinks) or >30 g per day for males (2.0 standard alcohol drinks) (a standard drink contains 14 g of alcohol: 12 oz of beer, 5 oz of wine or 1.5 oz of spirits) or drug abuse. (1.0 fluid oz (US) = 29.57 ml)
  6. Any other clinically significant medical condition, as determined by the Investigator. These clinically significant medical conditions include, but are not limited to, uncontrolled hypertension, NYHA class III or IV CHF, proliferative diabetic retinopathy and neuropathic symptoms that limit activities of daily living.
  7. Participation in another clinical trial and/or treatment received with any investigational agent within one month before the initial dose of study medication.
  8. Concomitant therapy with the following: (See Appendix G for List of Drug Trade Names)

     1. weight loss medications
     2. oral or injected hypoglycemics (metformin is allowed) or insulin
     3. oral, parenteral or inhaled steroids; nasal, topical ocular, intravitreal, and low to moderate potency topical steroids are allowed
     4. dihydropyridine calcium channel blockers (amlodipine, diltiazem and verapamil are allowed)
     5. H2 antagonists and proton pump inhibitors (liquid and tablet antacids are allowed)
     6. midazolam, triazolam, alprazolam, terfenadine, astemizole, digoxin, coumarin derivatives, phenytoin, rifampin, HIV protease inhibitors, spironolactone, aliskiren, erythromycin or clarithromycin, cyclosporine or tacrolimus
     7. Subjects currently taking lipid lowering medications may be enrolled if the Investigator determines that the subject does not have any conditions that preclude cessation of lipid lowering treatment for up to 12 weeks. [All subjects will be required to discontinue all lipid lowering therapies during the 4 week Pre-Treatment Period and will then be randomized to receive either atorvastatin 10 mg or atorvastatin placebo during the first 8 weeks of the Treatment Period. All subjects will then receive atorvastatin 10 mg during weeks 8 to 16 of the Treatment Period.] Subjects may not be on any other lipid lowering agent through Visit 7 (Week 20) of the study.
  9. History of HIV
  10. Positive hepatitis B (HbsAg) or positive hepatitis C (Hepatitis C antibody) test during Screening
  11. Liver function tests must not be above the following cut-offs: ALT and/or AST >3.0X ULN, AP >1.5X ULN and total bilirubin >ULN. (If all LFTs are WNL and total bilirubin is elevated, a retest of direct and indirect bilirubin may be performed. Subjects with indirect total bilirubin up to 3X ULN (presumed Gilbert's syndrome) may be enrolled if all other LFTs are WNL.)
  12. CK must not be >2.5X ULN if not clearly related to recent exercise, injury or unusual activity
  13. Creatinine must not be >1.4 mg/dl in females and >1.5 mg/dl in males.
  14. Thyroid stimulating hormone level >1.5X ULN
  15. History of lactic acidosis
  16. Known hypersensitivity to cosyntropin (ACTH) or any component of the formulation (mannitol or sodium chloride)
  17. Known intolerance to statin drugs
  18. Any other condition which increases the risk of participation in the trial in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-03 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
1. The primary efficacy endpoint will be change from baseline to the end of treatment (Study Visit 6, Week 16) in HbA1c | 16 weeks

SECONDARY OUTCOMES:
1. Change from baseline to Week 8 in total and LDL-cholesterol (LDL-C) 2. Change from baseline to the end of treatment (Week 16) in the following : Seated blood pressure (systolic, diastolic and mean arterial pressure) Fasting blood glucose | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sherwyn Schwartz, MD, Principal Investigator — Diabetes & Glandular Disease Research Associates
Locations (24):
- United States (12):
  - Dr. Terence Hart, Muscle Shoals, Alabama
  - Genova Research, Tucson, Arizona
  - Research Solutions, Jonesboro, Arkansas
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Advanced Medical Research, Lakewood, California
  - Mills-Peninsula Helath Services, San Mateo, California
  - Diabetes Research Goup University of Hawaii at Manoa, Honolulu, Hawaii
  - Creighton Diabetes Center, Omaha, Nebraska
  - AHS Oklahoma Physician Group, Tulsa, Oklahoma
  - Covance Clinical Research Unit - Dr. Andrew Ahmann, Portland, Oregon
  - Covance CRU, Austin, Texas
  - Diabetes Glandular and Disease Research Associates, San Antonio, Texas
- Australia (8):
  - Flinders Medical Centre, Adelaide, South Australia
  - Lyell McEwin Hospital, North Western Adelaide, South Australia
  - ECRU, Box Hill, Melbourne, Victoria
  - School of Medicine and Pharmacology, Fremantle, Western Australia
  - Keough Institute, Nedands, Western Australia
  - Endocrinology Research Unit, Herston Road
  - Endocrinology Department, St Leonards
  - Royal Melbourn Hospital, Victoria
- New Zealand (4):
  - Middlemore Hospital, Otahuhu, Auckland
  - Lipid and Diabetes Research, Christchurch
  - Waikaito Hospital, Hamilton
  - Diabetes Centre, Wellington